CLINICAL TRIAL: NCT03182465
Title: Predictive Value of ProCalcitonin for the Detection of Bacteraemia in Patients Presenting to the Emergency Department for Low Risk Chemo-induced Febrile Neutropenia According to the MASCC Score: a Prospective, Monocentric Observational Study (CALIF)
Brief Title: Predictive Value of ProCalcitonin for the Detection of Bacteraemia in Patients Presenting to the Emergency Department for Low Risk Chemo-induced Febrile Neutropenia
Acronym: CALIF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017/24FEV/112
Record Dates: First submitted 2017-06-08; First posted 2017-06-09 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Febrile Neutropenia, Drug-Induced
MeSH Terms: conditions — Chemotherapy-Induced Febrile Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the predictive value of ProCalcitonin (Other): Patients with solid tumors admitted at the emergency care presenting a febrile neutropenia due to chemotherapy
  Interventions: Diagnostic Test: Value of ProCalcitonin

INTERVENTIONS:
Diagnostic Test: Value of ProCalcitonin — The predictive value of ProCalcitonin in patients with solid tumors presenting a febrile neutropenia due to chemotherapy at emergency unit will be a factor to detect the level of bacteria.

SUMMARY:
CALIF study is a monocentric observational study which aim is to analyse the value of adding procalcitonin (PCT, a pre-hormon increased in bacterial infection and septicaemia) in the management of chemo-induced febrile neutropenia occurring in patient with solid tumour. Febrile neutropenia will be managed according to international guidelines. PCT will be dosed at initial presentation. Primary objective is to determine the optimal value of PCT for the detection of septicaemia in low risk (according to MASCC score). The investigators plan also to compare two risk stratification scores: the validated MASCC score and a recently developed score which includes PCT and other more objective items.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old
* Patients with solid malignant tumor treated by chemotherapy (neoadjuvant, concomittant, adjuvant or metastatic)
* Febrile neutropenia chemo-induced (fever > 38°C, neutrophils < 500 /microliter or nadir < 500 /microliter)
* Patients non hospitalized at the event (when he presented febrile neutropenia)
* Informed consent signed

Exclusion Criteria:

* Thyroid medullar carcinoma
* Patient not able to understand protocol (mental retardation, psychiatric disorders, .... )

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
Minimum level of ProCalcitonin | at day 0
  Bacteria detection will be determined by the optimal value of ProCalcitonin in patients with solid tumors treated by chemotherapy and at low MASCC risk

SECONDARY OUTCOMES:
Compare the MASCC score and the Anh & al score | up to 1 week
  Based on the chareteristics of the two scores

CONTACTS AND LOCATIONS:
Overall Officials: jean-Pascal Machiels, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan to share IPD at this moment